CLINICAL TRIAL: NCT01808209
Title: Clinical Performance of Stenfilcon A Versus Filcon II 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: EX-MKTG-40
Record Dates: First submitted 2013-02-14; First posted 2013-03-11 (Estimated); Results first posted 2015-01-19 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- stenfilcon A (Experimental): Participants wear a first pair of lenses for one week and then crossover and wear an alternate second pair of lenses for one week.
  Interventions: Device: filcon II 3
- filcon II 3 (Active Comparator): Participants wear a first pair of lenses for one week and then crossover and wear an alternate second pair of lenses for one week.
  Interventions: Device: stenfilcon A

INTERVENTIONS:
Device: stenfilcon A — Participants wear a first pair of lenses for one week and then crossover and wear an alternate second pair of lenses for one week.
  Other Names: stenfilcon A (Daily Disposable Contact Lens)
  Arms: filcon II 3
Device: filcon II 3 — Participants wear a first pair of lenses for one week and then crossover and wear an alternate second pair of lenses for one week.
  Other Names: filcon II 3 (Daily Disposable Contact Lens)
  Arms: stenfilcon A

SUMMARY:
Clinical Performance of Stenfilcon vs. Filcon II 3

DETAILED DESCRIPTION:
The objective of this study is to compare the comfort and clinical performance of Stenfilcon vs. Filcon II 3 compared to subject's habitual contact lenses. The null hypothesis is that there is no difference in the clinical performance between the two sets of lenses.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following conditions prior to inclusion in the study:

* Based on his/her knowledge, must be in good general health. Be of legal age (18 years) or older.
* Be able and willing to adhere to the instructions set forth in this protocol and complete all specified evaluation.
* Read, indicate understanding of, and sign Written Informed Consent (Appendix 1)
* Require a contact lens prescription between -0.50 and -6.00 and have no more than -.75dioptor (D) of astigmatism in both eyes
* Achieve visual acuity of 6/9 or better in each eye with a spherical contact lens prescription.
* An existing soft contact lens wearer of any modality.
* Must be able to wear their lenses at least 6 full days over the 7 days; 14 hours per day, assuming there are no contraindications for doing so.
* Have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having:
* No amblyopia.
* No evidence of lid abnormality or infection (e.g. entropion, ectropion, chalazia, recurrent styes).
* No clinically significant slit lamp findings (e.g. infiltrates or other slit lamp findings greater than Grade 2: corneal edema, tarsal abnormalities, and conjunctival injection).
* No other active ocular disease (e.g. glaucoma, history of recurrent corneal erosions, cornea [infiltrates], conjunctiva, lids, and intraocular infection or inflammation of an allergic, bacterial, or viral etiology.)
* No aphakia

Exclusion Criteria:

Any of the following will render a subject ineligible for inclusion:

* Neophytes, who have not worn lenses before
* Greater than 0.75D of refractive astigmatism in either eye
* Presence of clinically significant (grade 3 or above) anterior segment abnormalities; inflammations such as iritis; or any infection of the eye, lids, or associated structures.
* Presence of ocular or systemic disease or need of medication which might interfere with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear such as:
* Pathological dry eye or associated findings
* Pterygium, pinguecula or corneal scars within the visual axis
* Neovascularization > 0.75 mm in from the limbus
* Giant papillary conjunctivitis (GPC) Grade 3 or above
* Anterior uveitis or iritis (past or present)
* Seborrheic eczema, seborrheic conjunctivitis
* History of corneal ulcer or fungal infections
* Poor personal hygiene
* A known history of corneal hypoesthesia (reduced corneal sensitivity).
* Contact lens best corrected Snellen visual acuities (VA) worse than 6/9
* Aphakia, Keratoconus or a highly irregular cornea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Wolffsohn, PhD, Principal Investigator — University of Aston Birmingham, West Midlands, United Kingdom
Locations (1):
- University of Aston, Birmingham, West Midlands, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty habitual contact lens wearing subjects were recruited by the Optometry Clinic at Aston University
Pre-assignment Details: All subjects were habitual lens wearers and were randomized to each pair of study lenses. Only one patient failed to complete all study visits and their data was excluded from the analysis.
Groups:
- Stenfilcon A Then Filcon II 3: All participants completing the study were habitual lens wearers. All participants wore both sets of study lenses. Participants were randomized to wear either pair of study lenses as a first pair and then crossed over to wear the alternate second pair of study lenses. Each worn one week.
- Filcon II 3 Then Stenfilcon A: All participants completing the study were habitual lens wearers. All participants wore both sets of study lenses. Participants were randomized to wear either pair of study lenses as a first pair and then crossed over to wear the alternate second pair of study lenses. Each pair worn one week.
Period: Overall Study
Arm/Group | Stenfilcon A Then Filcon II 3 | Filcon II 3 Then Stenfilcon A
Started | 33 | 27
Completed | 33 | 26
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants completing the study wore both sets of study lenses.Participants were randomized to wear a first pair of lenses for one week and then crossover and wear an alternate second pair of lenses for one week.
Groups:
- Filcon II 3 Then Stenfilcon A: All participants completing the study were habitual lens wearers. All participants wore both sets of study lenses. Participants were randomized to wear either pair of study lenses as a first pair and then crossed over to wear the alternate second pair of study lenses. Each worn one week.
- Total: Total of all reporting groups
Arm/Group | Stenfilcon A Then Filcon II 3 | Filcon II 3 Then Stenfilcon A | Total
Number analyzed (Participants) | 33 | 26 | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 26 | 59
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 42
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United Kingdom | 33 | 26 | 59

OUTCOME MEASURES:

1. Primary Outcome: Daily and Comfortable Wearing Time
Description: Participant rating of lens Daily and Comfortable Wearing Time. Collected at baseline for all habitual lenses.(The hours of average comfortable wearing time and average daily wearing time.)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Overall Study Group: All 59 subjects with habitual lens prior to dispense of study lenses.
Arm/Group | Overall Study Group
Number analyzed (Participants) | 59
hours
  Average Wearing Time | 9.8 (3.1)
  Average Comfortable Wearing Time | 7.7 (3.4)

2. Primary Outcome: Daily and Comfortable Wearing Time
Description: Participant rating of lens Daily and Comfortable Wearing Time. Collected at 1 week wear for each lens.(The hours of average comfortable wearing time and average daily wearing time.)
Time Frame: 1 week
Population: All 59 subjects were habitual lens wearers and randomized to both sets of study lenses.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Stenfilcon A; Filcon II 3: All participants completing the study were habitual lens wearers. All participants wore both sets of study lenses. Participants were randomized to wear either pair of study lenses as a first pair and then crossed over to wear the alternate second pair of study lenses. Each worn one week.
Arm/Group | Stenfilcon A | Filcon II 3
Number analyzed (Participants) | 59 | 59
hours
  Average Wearing Time | 11.4 (2.6) | 10.8 (2.6)
  Average Comfortable Wearing Time | 8.7 (3.0) | 8.7 (2.8)

3. Primary Outcome: Handling
Description: Participant rating for lens handling. Collected at 1 week. (Insertion: 0-100, 0= could not get it in and 100= went in without a problem. Removal: 0= could not get it out and 100= came out without a problem. Blister: 0=impossible and 100=came out extremely easily).
Time Frame: 1 Week
Population: All 59 subjects were habitual lens wearers and randomized to both sets of study lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A | Filcon II 3
Number analyzed (Participants) | 59 | 59
units on a scale
  From Blister | 90.8 (11.7) | 92.2 (0.32)
  Inside Out | 84.9 (24.6) | 86.4 (25.9)
  Insertion | 93.4 (10.7) | 89.3 (13.0)
  Removal | 90.0 (13.6) | 92.0 (11.3)

4. Primary Outcome: Comfort
Description: Participant rating of lens comfort. Collected at baseline for habitual pair. (0-100; 0=very uncomfortable,100=extreme comfort / cannot feel them at all)
Time Frame: Baseline
Population: All 59 subjects were habitual lens wearers and randomized to both sets of study lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Habitual Lens: All participants completing the study were habitual lens wearers. All participants wore both sets of study lenses. Participants were randomized to wear either pair of study lenses as a first pair and then crossed over to wear the alternate second pair of study lenses. Each pair was worn one week.
Arm/Group | Habitual Lens
Number analyzed (Participants) | 59
units on a scale
  On Insertion | 85.0 (17.0)
  After 4 Hours | 91.8 (9.1)
  After 8 Hours | 80.8 (15.7)
  On Removal | 75.3 (19.7)

5. Primary Outcome: Comfort
Description: Participant rating for comfort. Collected at 1 week. (0-100, 0= very uncomfortable and 100= extreme comfort/cannot feel them at all).
Time Frame: 1 Week
Population: All 59 subjects were habitual lens wearers and randomized to both sets of study lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A | Filcon II 3
Number analyzed (Participants) | 59 | 59
units on a scale
  Insertion | 93.0 (9.6) | 90.6 (13.2)
  After 4 hours | 89.7 (14.6) | 88.8 (11.8)
  After 8 hours | 81.7 (17.7) | 79.0 (17.6)
  Removal | 75.8 (18.8) | 72.4 (20.0)

6. Primary Outcome: Dryness
Description: Participant rating of lens dryness. Collected at baseline for habitual pair. (0-100; 0=very uncomfortable, 100=extreme comfort/ cannot feel them at all)
Time Frame: Baseline
Population: All 59 subjects were habitual lens wearers and randomized to both sets of study lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Habitual Lens
Number analyzed (Participants) | 59
units on a scale
  On Insertion | 85.6 (26.8)
  After 4 Hours | 84.0 (21.7)
  After 8 Hours | 73.8 (22.0)
  On Removal | 67.1 (25.3)

7. Secondary Outcome: Blood Vessel Coverage
Description: Assessment of ocular health. Collected at baseline after removal of lenses. Percent of blood vessel coverage.
Time Frame: Baseline
Population: Prior to randomization
Measure: Mean (Standard Deviation); unit: percentage of blood vessel coverage
Units Other Than Participants: Eyes
Arm/Group | Overall Study Group
Number analyzed (Participants) | 59
Number analyzed (Eyes) | 118
percentage of blood vessel coverage
  Right Eye | 3.68 (3.05)
  Left Eye | 3.74 (2.74)

8. Primary Outcome: Dryness
Description: Participant rating for dryness. Collected at 1 week. (0-100, 0= very uncomfortable and 100= extreme comfort/cannot feel them at all).
Time Frame: 1 Week
Population: All 59 subjects were habitual lens wearers and randomized to both sets of study lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A | Filcon II 3
Number analyzed (Participants) | 33 | 26
units on a scale
  Insertion | 94.4 (11.8) | 93.6 (11.6)
  After 4 hours | 88.9 (13.3) | 88.0 (12.4)
  After 8 hours | 78.5 (19.0) | 79.2 (16.7)
  Removal | 72.9 (21.1) | 70.8 (19.1)

9. Primary Outcome: Vision Quality
Description: Participant rating of vision quality. Collected at baseline for habitual lens. (0-100; 0=extremely poor vision totally blurred 100=excellent vision totally sharp)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Study Group
Number analyzed (Participants) | 59
units on a scale | 92.2 (8.6)

10. Primary Outcome: Vision Quality
Description: Participant rating of vision quality. Collected at 1 week. (0-100; 0=extremely poor vision totally blurred 100=excellent vision totally sharp)
Time Frame: 1 Week
Population: All 59 subjects were habitual lens wearers and randomized to both sets of study lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A | Filcon II 3
Number analyzed (Participants) | 59 | 59
units on a scale | 89.9 (11.2) | 89.0 (11.7)

11. Primary Outcome: Eye Whiteness
Description: Participant rating for eye whiteness. Collected at baseline for habitual lenses. (0-100, 0= total redness and 100= totally white).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Study Group
Number analyzed (Participants) | 59
units on a scale | 82.5 (15.0)

12. Primary Outcome: Eye Whiteness
Description: as for outcome 11
Time Frame: 1 Week
Population: All 59 subjects were habitual lens wearers and randomized to both sets of study lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A | Filcon II 3
Number analyzed (Participants) | 59 | 59
units on a scale | 85.3 (12.5) | 84.9 (13.5)

13. Primary Outcome: Overall Satisfaction
Description: Participant rating for overall satisfaction. Collected at baseline for habitual lenses. (0-100, 0= extremely dissatisfied and 100= extremely satisfied).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Overall Study Group
Number analyzed (Participants) | 59
units on a scale | 88.1 (14.0)

14. Primary Outcome: Overall Satisfaction
Description: Participant rating for overall satisfaction. Collected at 1 week for study lenses. (0-100, 0= extremely dissatisfied and 100= extremely satisfied).
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Stenfilcon A | Filcon II 3
Number analyzed (Participants) | 59 | 59
units on a scale | 85.7 (12.4) | 82.5 (16.1)

15. Primary Outcome: Visual Acuity logMAR
Description: Assessment of Monocular (MHCVA) Right eye (OD), left eye (OS) and Binocular High Contrast Distance Visual Acuity (BHCVA). Collected at baseline for habitual lens. logMAR.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Overall Study Group
Number analyzed (Participants) | 59
logMAR
  MHCVA OD | -0.01 (0.08)
  MHCVA OS | -0.01 (0.08)
  BHCVA | -0.05 (0.07)

16. Primary Outcome: Visual Acuity logMAR
Description: Assessment of Monocular (MHCVA) Right eye (OD), left eye (OS) and Binocular High Contrast Distance Visual Acuity (BHCVA). Collected at dispense for study lenses. logMAR.
Time Frame: Dispense
Population: All 59 subjects were habitual lens wearers and randomized to both sets of study lenses.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Stenfilcon A | Filcon II 3
Number analyzed (Participants) | 59 | 59
logMAR
  MHCVA OD | -0.09 (0.10) | -0.07 (0.07)
  MHCVA OS | -0.09 (0.08) | -0.07 (0.06)
  BHCVA | -0.12 (0.08) | -0.11 (0.07)

17. Primary Outcome: Visual Acuity logMAR
Description: Assessment of Binocular High Contrast Distance Visual Acuity (BHCVA). Collected at 1 week for study lenses. logMAR
Time Frame: 1 Week
Population: All 59 subjects were habitual lens wearers and randomized to both sets of study lenses.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Stenfilcon A | Filcon II 3
Number analyzed (Participants) | 59 | 59
logMAR | -0.06 (0.06) | -0.03 (0.07)

18. Secondary Outcome: Blood Vessel Coverage
Description: Assessment of ocular health. Collected at 1 week after removal of lenses. Percentage of blood vessel coverage.
Time Frame: 1 Week
Population: All 59 subjects were habitual lens wearers and randomized to both sets of study lenses.
Measure: Mean (Standard Deviation); unit: percentage of blood vessel coverage
Units Other Than Participants: Eyes
Groups:
- Filcon II 3: All participants completing the study were habitual lens wearers. All participants wore both sets of study lenses. Participants were randomized to wear either pair of study lenses as a first pair and then crossed over to wear the alternate second pair of study lenses. Each pair worn one week.
Arm/Group | Stenfilcon A | Filcon II 3
Number analyzed (Participants) | 59 | 59
Number analyzed (Eyes) | 118 | 118
percentage of blood vessel coverage
  Right Eye | 4.63 (2.90) | 4.41 (2.94)
  Left Eye | 5.00 (3.32) | 5.25 (4.42)

19. Secondary Outcome: Conjunctival Redness
Description: Assessment of ocular health. Collected at baseline after removal of lenses. Percentage of conjunctival redness.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of redness
Units Other Than Participants: Eyes
Arm/Group | Overall Study Group
Number analyzed (Participants) | 59
Number analyzed (Eyes) | 118
percentage of redness
  Right Eye | 35.1 (1.0)
  Left Eye | 35.2 (1.2)

20. Secondary Outcome: Conjunctival Redness
Description: Assessment of ocular health. Collected at 1 week after removal of lenses. Percentage of conjunctival redness.
Time Frame: 1 Week
Population: All 59 subjects were habitual lens wearers and randomized to both sets of study lenses.
Measure: Mean (Standard Deviation); unit: percentage of redness
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A | Filcon II 3
Number analyzed (Participants) | 59 | 59
Number analyzed (Eyes) | 118 | 118
percentage of redness
  Right Eye | 35.6 (1.4) | 35.4 (1.3)
  Left Eye | 35.8 (1.4) | 35.4 (1.3)

21. Secondary Outcome: Corneal Staining
Description: Assessment of ocular health. Collected at baseline after removal of lenses. (Biomicroscopy, 0-4, 0=none , 4=severe )
Time Frame: Baseline
Population: Prior to randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Overall Study Group
Number analyzed (Participants) | 59
Number analyzed (Eyes) | 118
units on a scale | 0.6 (0.6)

22. Secondary Outcome: Corneal Staining
Description: Assessment of ocular health. Collected at 1 week after removal of lenses. (Biomicroscopy, 0-4, 0=none , 4=severe )
Time Frame: 1 Week
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A | Filcon II 3
Number analyzed (Participants) | 59 | 59
Number analyzed (Eyes) | 118 | 118
units on a scale | 0.4 (0.4) | 0.5 (0.4)

23. Secondary Outcome: Conjunctival Staining
Description: Assessment of ocular health. Collected at 1 week after removal of lenses. (Biomicroscopy, 0-4, 0=none , 4=severe )
Time Frame: 1 Week
Population: All 59 subjects were habitual lens wearers and randomized to both sets of study lenses.
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A | Filcon II 3
Number analyzed (Participants) | 59 | 59
Number analyzed (Eyes) | 118 | 118
units on a scale | 0.6 (0.5) | 0.6 (0.4)

24. Primary Outcome: Wettability
Description: Participant rating for surface wettability. Collected at 1 week. Tear film analysis in seconds.
Time Frame: 1 Week
Population: All 59 subjects were habitual lens wearers and randomized to both sets of study lenses.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Eyes
Arm/Group | Stenfilcon A | Filcon II 3
Number analyzed (Participants) | 59 | 59
Number analyzed (Eyes) | 118 | 118
seconds
  Right Eye | 10.9 (6.5) | 9.2 (5.4)
  Left Eye | 11.6 (9.0) | 9.6 (6.1)

ADVERSE EVENTS:
Time Frame: From dispense up to one week for each pair of lenses.
Groups:
- Stenfilcon A; Filcon II 3: All participants completing the study wore both sets of study lenses.Participants were randomized to wear a first pair of lenses for one week and then crossover and wear an alternate second pair of lenses for one week.
Arm/Group | Stenfilcon A | Filcon II 3
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigators will not be permitted to publish or present at scientific meetings results obtained from the clinical study without prior written consent from the sponsor. Assuming that the product is marketed, and only with the sponsor's permission, will they allow publication of the results of the study.